CLINICAL TRIAL: NCT04155073
Title: Development and Testing of an Electronic Visit for COPD Early Detection and Smoking Cessation
Brief Title: E-Visit for COPD and Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jennifer Dahne, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00086016
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Cigarette Smoking; Telemedicine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cigarette Smoking | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD/smoking cessation electronic visit (e-visit) (Experimental): This group will be sent 1) an invitation to complete an electronic visit (e-visit) focused on cigarette smoking, quitting smoking, and respiratory symptoms, 2) an invitation to complete a follow-up e-visit one-month after the initial e-visit, and if needed, 3) a home spirometry test with instructions on how to video themselves completing a lung functioning test via the device within an additional e-visit.
  Interventions: Behavioral: smoking cessation, early COPD detection, electronic visit
- Treatment as Usual (TAU) (Active Comparator): This group will be provided information about the state quitline and about the importance of quitting smoking and it will be recommended that they contact their PCP to schedule a medical visit to discuss quitting smoking.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: smoking cessation, early COPD detection, electronic visit — electronic visits (e-visits) for smoking cessation and early detection of chronic obstructive pulmonary disease (COPD)
  Arms: COPD/smoking cessation electronic visit (e-visit)
Other: Treatment As Usual — Information about the state quitline and about the importance of quitting smoking and a recommendation to contact one's PCP to schedule a medical visit to discuss quitting smoking
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this work is to develop, refine, and pilot test an electronic visit (e-visit) to: 1) deliver smoking cessation treatment to adults at risk for COPD and 2) to improve rates of COPD early detection and accurate diagnosis. The investigators will conduct a pilot RCT of the COPD/smoking cessation e-visit as compared to treatment as usual (TAU), with primary objective to provide effect size estimates for a larger RCT.

ELIGIBILITY:
Inclusion Criteria:

* current cigarette smoker,
* enrolled in MUSC's Epic MyChart program or willing to sign up for MyChart,
* possess a valid e-mail address that is checked daily,
* English fluency, and
* owner of an iOS or Android-compatible smartphone and a webcam-enabled device

Exclusion Criteria:

* COPD on a patient's problem list within Epic.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Dahne J, Player MS, Strange C, Carpenter MJ, Ford DW, King K, Miller S, Kruis R, Hawes E, Hidalgo JE, Diaz VA. Proactive Electronic Visits for Smoking Cessation and Chronic Obstructive Pulmonary Disease Screening in Primary Care: Randomized Controlled Trial of Feasibility, Acceptability, and Efficacy. J Med Internet Res. 2022 Aug 30;24(8):e38663. doi: 10.2196/38663. PMID 36040766

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COPD/Smoking Cessation Electronic Visit (E-visit) | Treatment as Usual (TAU)
Started | 85 | 40
Completed | 85 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COPD/Smoking Cessation Electronic Visit (E-visit) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 85 | 40 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.12 (9.75) | 51.93 (8.52) | 53.42 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 22 | 74
  Male | 33 | 18 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 83 | 38 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 9 | 27
  White | 59 | 28 | 87
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Evidence-based Cessation Treatment Utilization
Description: participants in both groups will be queried for use of a smoking cessation medication since the last assessment
Time Frame: Baseline through Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | COPD/Smoking Cessation Electronic Visit (E-visit) | Treatment as Usual (TAU)
Number analyzed (Participants) | 85 | 40
Participants
  Month 1 | 44 | 10
  Month 3 | 51 | 11

2. Primary Outcome: Number of Participants at Month 1 and Month 3 With At Least 1 Quit Attempt
Description: quit attempts will be assessed at each follow-up using a timeline followback for the last 6-months at baseline and since prior follow-up for each subsequent assessment
Time Frame: Baseline through Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | COPD/Smoking Cessation Electronic Visit (E-visit) | Treatment as Usual (TAU)
Number analyzed (Participants) | 85 | 40
Participants
  Month 1 | 20 | 6
  Month 3 | 24 | 13

3. Secondary Outcome: E-visit Acceptability and Feasibility
Description: the percentage of patients who complete the initial and follow-up e-visits
Time Frame: Baseline through Month 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | COPD/Smoking Cessation Electronic Visit (E-visit) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/40
Other Adverse Events (participants affected / at risk) | 0/85 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT04155073/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04155073/ICF_002.pdf